CLINICAL TRIAL: NCT02537483
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group, Clinical Study Comparing the Efficacy and Safety of IDP-120 Gel in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing the Efficacy and Safety of IDP-120 Gel in the Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valeant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-120A-201
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDP-120 Gel (Experimental): IDP-120 Gel, applied topically to the face once daily for 12 weeks.
  Interventions: Drug: IDP-120 Gel
- IDP-120 Component A (Active Comparator): IDP-120 Component A, applied topically to the face once daily for 12 weeks
  Interventions: Drug: IDP-120 Component A
- IDP-120 Component B (Active Comparator): IDP-120 Component B, applied topically to the face once daily for 12 weeks
  Interventions: Drug: IDP-120 Component B
- IDP-120 Vehicle Gel (Placebo Comparator): IDP-120 Vehicle Gel, applied topically to the face once daily for 12 weeks
  Interventions: Drug: IDP-120 Vehicle Gel

INTERVENTIONS:
Drug: IDP-120 Gel — Investigational Product: IDP-120 Gel
  Arms: IDP-120 Gel
Drug: IDP-120 Component A — Comparator Product: IDP-120 Component A
  Arms: IDP-120 Component A
Drug: IDP-120 Component B — Comparator Product: IDP-120 Component B
  Arms: IDP-120 Component B
Drug: IDP-120 Vehicle Gel — Comparator Product: IDP-120 Vehicle Lotion
  Arms: IDP-120 Vehicle Gel

SUMMARY:
The primary objective of this study is to compare the efficacy, safety, and tolerability of IDP-120 Gel to IDP-120 Component A, IDP-120 Component B, and IDP-120 Vehicle Gel in subjects with moderate to severe acne vulgaris.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, tolerability, and efficacy of IDP-120 Gel in comparison with IDP-120 Component A, IDP-120 Component B, and IDP-120 Vehicle Gel at Weeks 2, 4, 8, and 12 in subjects with moderate to severe acne. IDP-120 is a gel for the topical treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 9 years of age and older
* Written and verbal informed consent must be obtained.
* Subject must have a score of moderate or severe on the Evaluator's Global Severity assessment at the screening and baseline visit
* Pre-menses females and women of childbearing potential must have a negative urine pregnancy test at screening and baseline visits
* Subjects must be willing to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

* Any dermatological conditions on the face that could interfere with clinical evaluations
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive
* Subjects with a facial beard or mustache that could interfere with the study assessments
* Subjects who are unable to communicate or cooperate with the Investigator
* Subjects with any underlying disease that the Investigator deems uncontrolled and poses a concern for the subject's safety while participating in the study

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Absolute change from Baseline to Week 12 in mean inflammatory lesion counts | 12 weeks
  At each visit the Evaluator will count the total number of inflammatory lesions (papules, pustules, and nodules) on the subject's face.
  Inflammatory lesions are defined as follows:
  Papule - a small, solid elevation less than 5 mm in diameter. Most of the lesion is above the surface of the skin.
  Pustule - a small, circumscribed elevation less than 5 mm in diameter that contains yellow-white exudate.
  Nodule - a subcutaneous lesion greater than or equal to 5 mm in diameter.
Absolute change from Baseline to Week 12 in mean non-inflammatory lesion counts | 12 weeks
  At each visit the Evaluator will count the total number of non-inflammatory lesions (open and closed comedones).
  Non-inflammatory lesions are defined as follows:
  Open comedones (black head) - a lesion in which the follicle opening is widely dilated with the contents protruding out onto the surface of the skin.
  Closed comedones (white head)- a lesion in which the follicle opening is closed, but the sebaceous gland is enlarged by the pressure of the sebum build up, which in turn causes the skin around the follicle to thin and become elevated with a white appearance.
Percent of subjects who achieve at least a two-grade reduction from baseline and are Clear or Almost Clear at Week 12 in the Evaluator's Global Severity Score. | 12 weeks
  At each visit the severity will be determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations will be scored on a scale of 0-4 (Evaluator's Global Severity Score), with 0 being clear and 4 being severe. Please see below for complete definitions.
  0. Clear - Normal, clear skin with no evidence of acne vulgaris
  1. Almost clear- Rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red)
  2. Mild- Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulo-cystic lesions)
  3. Moderate-Non-inflammatory lesions predominate, with multiple inflammatory lesions evident: several to many comedones and papules/pustules, and there may or may not be one nodulo-cystic lesion
  4. Severe- Inflammatory lesions are more apparent, many comedones and papules/pustules, there may or may not be up to 2 nodulo-cystic lesions.

SECONDARY OUTCOMES:
Absolute change in inflammatory and non-inflammatory lesion counts from baseline at Weeks 2, 4, and 8. | 2, 4, and 8 weeks
  At each visit the Evaluator will count the total number of inflammatory (papules, pustules, and nodules) and non-inflammatory (open and closed comedones) lesions on the subject's face, and the change will be calculated.
Percent of subjects who achieve at least a two-grade reduction from baseline and are Clear or Almost Clear at Week 2, 4, and 8 in the Evaluator's Global Severity Score | 2, 4, and 8 weeks
  At each visit the severity will be determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations will be scored on a scale of 0-4 (Evaluator's Global Severity Score), with 0 being clear and 4 being severe. Please see below for complete definitions.
  0. Clear - Normal, clear skin with no evidence of acne vulgaris
  1. Almost clear- Rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red)
  2. Mild- Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulo-cystic lesions)
  3. Moderate-Non-inflammatory lesions predominate, with multiple inflammatory lesions evident: several to many comedones and papules/pustules, and there may or may not be one nodulo-cystic lesion
  4. Severe- Inflammatory lesions are more apparent, many comedones and papules/pustules, there may or may not be up to 2 nodulo-cystic lesions.
Mean percent change in inflammatory and non-inflammatory lesion counts form baseline at Weeks 2, 4, 8, and 12. | 2, 4, 8, and 12 weeks
  At each visit the Evaluator will count the total number of inflammatory (papules, pustules, and nodules) and non-inflammatory (open and closed comedones) lesions on the subject's face, and the percent change will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, MS, Study Director — Valeant Pharmaceuticals